CLINICAL TRIAL: NCT04970836
Title: The Immune Responses After Hepatitis B Revaccination Doses in a Young Cohort
Acronym: IRHBRVD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Academia Sinica, Taiwan (Other); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202012221MINB; 110-2314-B-002-132 (Other Grant/Funding Number: The Ministry of Science and Technology)
Record Dates: First submitted 2021-07-06; First posted 2021-07-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis B; Vaccination; Infection; Preventable Disease, Vaccine
Keywords: hepatitis B vaccine; revaccination; young adult; booster
MeSH Terms: conditions — Hepatitis B; Infections; Vaccine-Preventable Diseases | interventions — Hepatitis B Vaccines; Engerix-B

STUDY DESIGN:
Intervention Model Description: prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low titer with two doses of HB Vaccines (Experimental): anti-HBs titer 2.5-10 mIU/mL with two doses of HB Vaccines at Day 0 and Day 28
  Interventions: Biological: recombinant hepatitis B vaccine
- Low titer with one dose of HB Vaccine (Active Comparator): anti-HBs titer 2.5-10 mIU/mL with one dose of HB Vaccine at Day 0
  Interventions: Biological: recombinant hepatitis B vaccine
- Extremely low titer with two doses of HB Vaccines (Active Comparator): anti-HBs titer lower than 2.5 mIU/mL with two doses of HB Vaccines at Day 0 and Day 28
  Interventions: Biological: recombinant hepatitis B vaccine
- Extremely low titer with one dose of HB Vaccine (Active Comparator): anti-HBs titer lower than 2.5 mIU/mL with one dose of HB Vaccine at Day 0
  Interventions: Biological: recombinant hepatitis B vaccine

INTERVENTIONS:
Biological: recombinant hepatitis B vaccine — Hepatitis B vaccine (Engerix-B) will be administered to the eligible participants by 4 groups. Each case will be tracked for 12 months, at 0, 7-10 days, 28 days, 24-28 weeks, 48-52 weeks anti-HBs titer concentration and 4 follow-up questionnaires.
  Other Names: Engerix-B

SUMMARY:
This prospective cohort study aims to provide the evidence-based clinical guide to help decide the revaccination doses of hepatitis B vaccine that the high-risk young adults without hepatitis B seroprotective antibodies (anti-HBs titer<10 mIU/mL) need to take.

DETAILED DESCRIPTION:
Purpose For young adults born after the neonatal hepatitis B immunization program, especially those who were 20-33 years old after 1987, additional hepatitis B vaccination may have the benefit of strengthening protection from acute hepatitis B infection among high-risk groups. However, how many doses are most appropriate for the protection of high-risk groups is still an issue to be resolved. This study aims to provide the evidence-based clinical guide to help decide the revaccination doses of hepatitis B vaccine that the high-risk young adults without hepatitis B seroprotective antibodies (anti-HBs titer<10 mIU/mL) need to take.

Materials and Methods From August 2021 to July 2024, the investigator will invite young adults born in Taiwan over the age of 20 and born after 1987, who have received a full course of hepatitis B vaccine at least three doses at their infant period. Those who are all negative for hepatitis B surface antibodies (anti-HBs) and surface antigens (HBsAg) are enrolled to 4 groups according to the anti-HBs titer concentration (anti-HBs titer between 2.5-10 mIU/mL is a low concentration, anti-HB titer less than 2.5 mIU/mL is an extreme low concentration) with one or two doses of hepatitis B vaccine (Engerix-B) administered, respectively. Each group recruits 60 cases to reach a total of 240 participants. Each participant was followed for 12 months, and the anti-HBs titer concentration was measured in 0, 7-10 days, 28 days, 24- 28 weeks, and 48-52 weeks. The investigator will calculate the anti-HBs titer reaction rate and immune response after receiving hepatitis B vaccine(s) at each stage, and do further univariate and multivariate analysis.

Expected Results This prospective cohort study can help understand the difference in the anti-HBs titer response after 1 or 2 revaccination doses by the anti-HBs titer concentration as well as the two different types of hepatitis B vaccination in childhood It is expected to provide an important reference for the administration of hepatitis B vaccine in young adults of high-risk groups.

ELIGIBILITY:
Inclusion Criteria:

1. The actual age at the time of admission was higher than 20 years old and birth year after 1987
2. Born in Taiwan and had received a full course of hepatitis B vaccines at least three doses at infant period.
3. Those who have tested negative for hepatitis B surface antibody and surface antigen at baseline
4. Have never been vaccinated against hepatitis B in childhood and adolescence by questionnaire
5. Consent to administer 1-2 doses of hepatitis B vaccine according to the assigned group after sharing decision making process
6. In good health

Exclusion Criteria:

1. Those who were previously allergic to hepatitis B vaccine or its components (such as yeast)
2. Those who have been vaccinated against hepatitis B during childhood and adolescence
3. Those who have a positive test for hepatitis B surface antibody or a positive test for hepatitis B surface antigen

Ages: 20 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
anti-HBs titer response rate at 7-10 days | 7-10 days
  the anti-HBs titer response rate after 1-2 doses of hepatitis B vaccine(s)
anti-HBs titer response rate at one month | 28 days
  the anti-HBs titer response rate after 1-2 doses of hepatitis B vaccine(s)
anti-HBs titer response rate at 6 months | 24-28 weeks
  the anti-HBs titer response rate after 1-2 doses of hepatitis B vaccine(s)
anti-HBs titer response rate at 12 months | 48-52 weeks
  the anti-HBs titer response rate after 1-2 doses of hepatitis B vaccine(s)
anti-HBs titer immune response change at 12 months | 48-52 weeks
  anti-HBs titer immune response change at 12 months after 1-2 doses of hepatitis B vaccine(s)

CONTACTS AND LOCATIONS:
Overall Officials: CHYI-FENG JAN, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Family Medicine, NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No